CLINICAL TRIAL: NCT03519490
Title: Myopia Progression in Children Wearing Near Center and Distance Center Multifocals - a Randomized Controlled Clinical Trial
Brief Title: Can Distance Center and Near Center Multifocal Contact Lenses Control Myopia Progression in Children?
Acronym: ADPADP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of interest and support
Sponsor: Thomas A. Aller, OD (Other)
Collaborators: SynergEyes, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Thomas A. Aller, OD, Principal Investigator, Aller, Thomas A., OD
Organization: Aller, Thomas A., OD (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SY-001001
Record Dates: First submitted 2018-04-17; First posted 2018-05-09 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Myopia; Myopia, Progressive
Keywords: Myopia; Myopia Control; Bifocal Contact Lenses; Multifocal Contact Lenses; Hybrid Contact Lenses; Randomized Controlled Clinical Trial; Distance Center Multifocal Contact Lens; Near Center Multifocal Contact Lens
MeSH Terms: conditions — Myopia; Myopia, Degenerative

STUDY DESIGN:
Intervention Model Description: Using a covariate adaptive randomization strategy, participants will be assigned to wear either multifocal or single vision Duette hybrid contact lenses for a period of two years. Additionally, subjects wearing the MFCLs will wear distance center in one eye and near center in the other eye, switching every six months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All lenses are identical in size, color and fitting characteristics. Lenses are supplied from the manufacturer with labels with full parameter information. This information will be removed or masked on the vials prior to being delivered to the office by the study coordinator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Single Vision Hybrid Contact Lens (Placebo Comparator): Subjects will wear the Duette single vision hybrid contact lens.
  Interventions: Device: Hybrid Contact Lens
- Multifocal Hybrid Contact Lens (Experimental): Subjects will wear the Duette hybrid multifocal contact lens with the near center design in one eye and the distance center design in the other eye with a crossover at every six months.
  Interventions: Device: Hybrid Contact Lens

INTERVENTIONS:
Device: Hybrid Contact Lens — Hybrid Single Vision or Multifocal Contact Lenses in Near Center and Distance Center Designs

SUMMARY:
Myopia has been increasing in prevalence and severity throughout the world over the last 30 years. Increasing levels of myopia are associated with increased frequency and severity of various ocular pathologies. Slowing myopia progression may help to reduce the future risks of these ocular pathologies.

Conventional spectacles and contact lenses correct myopia by moving the central focus of the eye from in front of the retina to on the retina centrally. To varying degrees, these lenses allow the light to focus behind the retina, at varying peripheral retinal locations. These findings have led to efforts to design spectacle and contact lenses which correct peripheral hyperopic defocus, to reduce myopia progression.

The consensus theory for how both multifocal contact lenses (MFCLs) and orthokeratology can control myopia progression is that they reduce, eliminate, or reverse relative peripheral hyperopic defocus. Existing published studies on the use of multifocal contact lenses to control myopia in humans have utilized lenses with the distance correction in the center with peripheral plus power to correct the peripheral blur.

It is possible that one of the mechanisms responsible for myopia progression control with MFCLs is that when the eye is exposed to an image focused on the retina and simultaneously an image anterior to the retina, that this will suppress axial elongation and myopia progression. This mechanism would not be dependent on whether the anterior image is located in the central area of the retina or the peripheral area of the retina. While there are no published human studies demonstrating the effectiveness of near center MFCLs, this author has presented retrospective data showing no differences in myopia progression between near center and distance center MFCLs.

Synergeyes, Inc.'s Duette contact lenses are hybrids of rigid gas permeable (RGP) with a silicon hydrogel peripheral portion or "skirt." They now make their MFCLs in both distance center (DC) and near center (NC) designs.

This study will analyze the myopia progression of children after being randomly assigned to wear Duette MFCLs or Duette standard single vision contact lenses over a span of two years. Subjects assigned to the MFCL group will wear a DC lens on one eye and a NC lens on the other and will reverse this lens assignment every six months. Refractive changes will be measured by cycloplegic autorefraction and axial lengths will be measured with a laser interference biometer (Zeiss IOLMaster) at six-month intervals.

DETAILED DESCRIPTION:
Nature & Purpose Myopia is the focus of growing attention and concern because of the now extremely high prevalence of myopia in some East Asian populations. For example, myopia prevalence figures in the low to mid 90's have been reported in some studies of University student populations in Taiwan and Shanghai, with a figure of 96.5% being reported for young adult Korean male conscripts in Seoul. Equivalent prevalence figures for the US have also been trending upwards, albeit lagging behind those of East Asia. For example, comparison of data from two studies of the same population over the time periods 1971-72 and 1999-2004, reveals an increase in the prevalence of myopia from 25% to 41.6% for the 12-54 year age range. These figures would not be of concern, were it not for the well-established link between myopia and sight-threatening ocular pathologies. Importantly, and as well summarized in a recent review by Ian Flitcroft, even low myopia is associated with an increased risk of pathology, with the latter, measured in terms of odds ratios, simply increasing with increasing myopia. Myopes are at increased risk of myopic maculopathy, retinal detachment, cataracts and glaucoma, with myopic maculopathy now the leading cause of monocular blindness in Japan and of new cases of blindness in Shanghai.

The rapidly changing myopia prevalence figures are consistent with the increasing acceptance of the role that environmental influences play in the development of myopia. Some but not all studies have linked myopia with increased near work, e.g., books read,8 and one recent German study showed a correlation between years of formal education with level of myopia. There are other studies pointing to outdoor activities being protective against the development of myopia. While unresolved are the specific factors contributing to myopia development and progression, that visual experience appears to play a central role has refocused attention on the possibility that myopia progression can and should be controlled.

Studies involving animal models for myopia (chicks, guinea pigs, marmosets, rhesus monkeys), provide compelling evidence for active emmetropization and a role for optical defocus in ocular growth modulation. Specifically, hyperopic defocus imposed on young eyes accelerates eye growth while imposed myopia slows it. Local retinal mechanisms have been implicated, with the peripheral retina apparently playing an important role in ocular growth regulation. Of relevance to the current study, in recent animal model studies, multifocal lenses incorporating zones of positive power were found to inhibit eye growth, even when these zones are limited to the periphery of the lenses. For already myopic eyes, both stabilization of myopia and reversal have been described.

The above observations with animal models, translated to human myopia, raise the possibility of increased progression with standard corrective spectacle and soft contact lenses, given that the image shell providing accurate on-axis focus typically falls increasingly behind the retina with increasing distance off-axis. Furthermore, more prolate eye shapes, a common finding in myopia, are expected to exaggerate this problem. Conversely, prescribing optical devices that impose peripheral myopic defocus are predicted to slow myopia progression, consistent with results from a number of independent myopia control studies involving orthokeratology, which produces a relative myopic shift in peripheral retinal defocus, a consequence of induced corneal shape changes.

While there are now many studies showing an average of around 50% control with both multifocal contact lenses and with orthokeratology, there are no published studies using either RGP or hybrid multifocal lenses for control of myopia. There are also no studies testing the efficacy of near center contact lenses for myopia control although animal studies suggest that the retinal location of imposed myopic defocus (i.e. focal plane in front of the retina), may not be critical to myopia control. Indeed, inhibited eye growth has been reported with positive adds located centrally, peripherally or in a multi-zonal format yet among clinicians there is a general belief that only multifocal contact lenses with peripheral adds work, no doubt a testament to the widely publicized finding in monkeys by Prof. Earl Smith's research group, that eye growth can be regulated by the peripheral retina alone. Nonetheless, Prof. Smith never stated that one could control myopia only through manipulation of the peripheral optics and indeed, his group more recently reported robust inhibitory effects on eye growth of multi-zonal lenses in monkeys.

The specific aim of this proposal is:

To compare the efficacy and thus merits of distance center and near center design bifocal hybrid contact lenses for controlling (slowing) progression of myopia in children and adolescents. Bifocal contact lens wearing participants will wear a distance center lens on one eye and a near center lens in their other eye, with one third of the participants wearing single vision contact lenses as a control (reference) group.

Outcome measures to be used to assess efficacy in the study include ocular refractions, corneal curvature and eye length at intervals, with data to be collected at 6 months intervals over a period of 24 months.

Participants Two groups of participants (all myopic), between the ages of 7 and 14 yr. (n=20 in the control group and n=40 in the test group), will be recruited. All will be fitted with either Duette single vision or bifocal contact lenses.

To be accepted into the study, participants will also need to be deemed suitable candidates for hybrid contact lenses. Successful single vision soft contact lens wearers will be automatically accepted into the study, while non-contact lens wearers will first undergo routine clinical pre-fitting assessment to verify their suitability for contact lens wear. To avoid excessive dropouts, only those who can demonstrate an ability to properly insert, remove and care for hybrid lenses will be enrolled.

Participants will be randomly assigned to each treatment group, i.e. single vision vs. bifocal hybrid contact lenses. To lessen the chance of a poorly randomized sample due to the small sample size, a modified covariate adaptive randomization method will be used.

Procedures All measurements specific to the vision screening, contact lens fitting and monitoring of myopia progression will be carried out at Thomas Aller's practice in San Bruno.

Once the participants have passed the screening protocol and read and signed the informed consent form, they will be required to attend a maximum of 10 office visits:

1. A baseline measurement session (this may be combined with screening and/or session 2)
2. A contact lens fitting session
3. A contact lens dispensing/training session
4. A routine contact lens follow-up session to verify that the lenses fit satisfactorily, and the lenses are not adversely affecting eye health
5. A 6-month follow-up measurement session
6. A 12-month follow-up measurement session
7. An 18-month follow-up measurement session
8. A 24-month follow-up measurement session.

The contact lens fitting session: Each participant will have their initial lenses selected, both single vision and bifocal lenses, based on the manufacturer's suggested fitting protocol. For all participants prescriptions will be modified as necessary to provide optimal distance vision, through both types of lenses (single vision and bifocal). Visual acuity will need to be at least 20/30 in the worse eye and at least 20/25 binocularly. Bifocal contact lens prescriptions will be selected to achieve both good distance and near vision. The add powers will be selected as the highest add power which results in acceptable distance visual acuity. The DCMF design allows for altering the zone sizes, but the default zone sizes will be used, subject to alteration as necessary to achieve good distance visual acuity. After Dr. Aller has determined the provisional prescriptions, the actual lens assignments will be made by a masked assistant. In this way it will be possible to mask and randomize the lens assignments appropriately. Bifocal contact lens wearers will also be randomly assigned to wear a distance center multifocal (DCMF) in one eye with the other eye wearing a near center multifocal (NCMF). At each six-month interval, the lens types assigned to the right and left eyes will be switched. The same procedure will be utilized for the single vision wearers, though this will only be a sham switch to help maintain masking. This crossover study design will help to identify any differences in myopia control efficacy between NC and DC designs, and also to lessen the chance of induced anisometropia, should there prove to be a difference in myopia control efficacy in these designs.

Follow-up contact lens review (aftercare) session: In order to verify that the lenses dispensed to the participants are fitting well and there are no complications regarding vision or the health of the eye, the participants will return for a follow-up appointment 2 weeks after the lenses have been dispensed. This is routine in clinical practice.

Follow-up visits at 6-month intervals: Baseline measurements will be repeated at the 6-month follow-up session (see Table 1 for measurements and procedures). The fit of the contact lenses and health of the front surface of the eye will be assessed also, as per routine contact lens practice. Adjustments to contact lens prescriptions may also be ordered, based on the results of this exam. If the prescription has changed by ≥ 0.5D or if the visual acuity has dropped below 20/30 in the worse eye or below 20/25 binocularly.

24-month follow-up measurement & aftercare session: Final measurements will be taken at this visit, repeating all baseline measurements. To lessen topographical changes induced by the rigid portion of the hybrid contact lenses, no lenses will be worn for 3 days prior to this visit.

Benefits In addition to the 3 comprehensive eye examinations received at no cost each participant will receive two years' supply of lenses and lens-related solutions. Professional fees for contact lens fittings and followup exams will be charged to the subjects at the standard rate for the practice. Also, through participation in this study, individuals will have the opportunity to learn more about their myopia and the overall health of their eyes. Finally if, at the end of the study, results show that a participant may benefit from the alternative treatment (single vision contact lenses vs. bifocal lenses), the participant will be informed and offered a prescription for the alternative treatment.

Risks The risks are limited to those associated with routine clinical procedures and are negligible. Reactions to local anesthetics are a rare but possible side-effect of their use for cycloplegia. Appropriate questioning of subjects and/or their parents about their prior experience with, and reaction to, local anesthetics, and exclusion of those with a history of previous reactions to local anesthetics can minimize this risk. Such reactions are treated with topical antibiotics and/or artificial tears and generally resolve within 24 hr. Hybrid contact lenses of both types are widely prescribed in routine clinical practice and the risks associated with their daily wear are minimal, given appropriate patient education and appropriately-timed "aftercare" exams. Aftercare exams are scheduled at 2 weeks, 6 and 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Myopia: ≥ 0.5 D in least myopic meridian, < 12.0 D in most myopic meridian);
* Anisometropia (interocular difference in refractive error) ≤ 2D
* Astigmatism: ≤ 3D
* Myopia progression ≥ 0.5D in at least one eye based on available clinical records or based on habitual spectacle prescription
* Visual acuity: best corrected acuity of 20/20 or better in each eye
* Capable of proper handling, insertion and removal of hybrid contact lenses

Exclusion Criteria:

* Ocular health: any pathology that may alter eye growth (e.g. history of retinal detachment & treatment for the same), and/or may adversely impact contact lens wear (e.g. chronic, poorly controlled allergic conjunctivitis) will be grounds for exclusion;
* Strabismus, amblyopia
* Systemic disease that may affect vision, vision development or contact lens wear
* Chronic use of medications that may affect immunity, such as oral or topical corticosteroids
* rigid or hybrid contact lens wear within the preceding 3 months;
* prior ocular surgery,
* nursing or pregnant mothers
* participants who cannot commit to the 24 month study period or who have a high likelihood of leaving the area within the 24 month study period

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Myopia progression rate | Data will be collected at baseline, that is to say at the beginning of the 24 month study, and also at six months after baseline, at 12 months, at 18 months and at study completion or 24 months.
  Change in myopia over time, expressed in terms of an annualized rate, based on cycloplegic spherical equivalent refractive error as measured by autorefraction.
Axial elongation rate | Data will be collected at baseline, that is to say at the beginning of the 24 month study, and also at six months after baseline, at 12 months, at 18 months and at study completion or 24 months.
  Change in axial length over time, expressed in terms of an annualized rate, based on measurement with the Zeiss IOLMaster.

SECONDARY OUTCOMES:
Subjective myopia progression rate | Data will be collected at baseline, that is to say at the beginning of the 24 month study, and also at six months after baseline, at 12 months, at 18 months and at study completion or 24 months.
  Change in myopia over time, expressed in terms of an annualized rate, based on cycloplegic spherical equivalent refractive error as measured by subjective refraction.
Macular Pigment Optical Density | Data will be collected at baseline and at 24 months from baseline at study completion.
  Macular pigment optical density is measured by the QuantifEye device.
Tear Film Dynamics and Meibomian Gland Health | Data will be collected at baseline and at 24 months from baseline at study completion.
  Lipid layer thickness, blink dynamics and meibomian gland health will be assessed with the Tear Science (Johnson & Johnson) Lipiview device.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Aller, OD, Principal Investigator
Locations (1):
- Dr. Thomas Aller Optometrist, Inc., San Bruno, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aller T, Wildsoet C. Optical control of myopia has come of age: or has it? Optom Vis Sci. 2013 May;90(5):e135-7. doi: 10.1097/OPX.0b013e31828b47cf. PMID 23528448
- [Background] Aller TA, Wildsoet C. Bifocal soft contact lenses as a possible myopia control treatment: a case report involving identical twins. Clin Exp Optom. 2008 Jul;91(4):394-9. doi: 10.1111/j.1444-0938.2007.00230.x. PMID 18601670
- [Background] Aller TA. Clinical management of progressive myopia. Eye (Lond). 2014 Feb;28(2):147-53. doi: 10.1038/eye.2013.259. Epub 2013 Dec 20. PMID 24357844
- [Background] Aller TA, Liu M, Wildsoet CF. Myopia Control with Bifocal Contact Lenses: A Randomized Clinical Trial. Optom Vis Sci. 2016 Apr;93(4):344-52. doi: 10.1097/OPX.0000000000000808. PMID 26784710
- [Background] Anstice NS, Phillips JR. Effect of dual-focus soft contact lens wear on axial myopia progression in children. Ophthalmology. 2011 Jun;118(6):1152-61. doi: 10.1016/j.ophtha.2010.10.035. Epub 2011 Jan 26. PMID 21276616
- [Background] Benavente-Perez A, Nour A, Troilo D. The effect of simultaneous negative and positive defocus on eye growth and development of refractive state in marmosets. Invest Ophthalmol Vis Sci. 2012 Sep 21;53(10):6479-87. doi: 10.1167/iovs.12-9822. PMID 22918633
- [Background] Arumugam B, Hung LF, To CH, Holden B, Smith EL 3rd. The effects of simultaneous dual focus lenses on refractive development in infant monkeys. Invest Ophthalmol Vis Sci. 2014 Oct 16;55(11):7423-32. doi: 10.1167/iovs.14-14250. PMID 25324283
- [Background] Benavente-Perez A, Nour A, Troilo D. Axial eye growth and refractive error development can be modified by exposing the peripheral retina to relative myopic or hyperopic defocus. Invest Ophthalmol Vis Sci. 2014 Sep 4;55(10):6765-73. doi: 10.1167/iovs.14-14524. PMID 25190657
- [Background] Berntsen DA, Kramer CE. Peripheral defocus with spherical and multifocal soft contact lenses. Optom Vis Sci. 2013 Nov;90(11):1215-24. doi: 10.1097/OPX.0000000000000066. PMID 24076542
- [Background] Chakraborty R, Read SA, Collins MJ. Hyperopic defocus and diurnal changes in human choroid and axial length. Optom Vis Sci. 2013 Nov;90(11):1187-98. doi: 10.1097/OPX.0000000000000035. PMID 24061153
- [Background] Cui Y, Li L, Wu Q, Zhao J, Chu H, Yu G, Wei W. Myopia correction in children: a meta-analysis. Clin Invest Med. 2017 Jun 26;40(3):E117-E126. doi: 10.25011/cim.v40i3.28391. PMID 28653613
- [Background] Fedtke C, Ehrmann K, Thomas V, Bakaraju RC. Peripheral Refraction and Aberration Profiles with Multifocal Lenses. Optom Vis Sci. 2017 Sep;94(9):876-885. doi: 10.1097/OPX.0000000000001112. PMID 28816867
- [Background] Holden B, Sankaridurg P, Smith E, Aller T, Jong M, He M. Myopia, an underrated global challenge to vision: where the current data takes us on myopia control. Eye (Lond). 2014 Feb;28(2):142-6. doi: 10.1038/eye.2013.256. Epub 2013 Dec 20. PMID 24357836
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Background] Huang J, Wen D, Wang Q, McAlinden C, Flitcroft I, Chen H, Saw SM, Chen H, Bao F, Zhao Y, Hu L, Li X, Gao R, Lu W, Du Y, Jinag Z, Yu A, Lian H, Jiang Q, Yu Y, Qu J. Efficacy Comparison of 16 Interventions for Myopia Control in Children: A Network Meta-analysis. Ophthalmology. 2016 Apr;123(4):697-708. doi: 10.1016/j.ophtha.2015.11.010. Epub 2016 Jan 27. PMID 26826749
- [Background] Jong M, Sankaridurg P, Li W, Resnikoff S, Naidoo K, He M. Reduced vision in highly myopic eyes without ocular pathology: the ZOC-BHVI high myopia study. Clin Exp Optom. 2018 Jan;101(1):77-83. doi: 10.1111/cxo.12563. Epub 2017 Jul 11. PMID 28696042
- [Background] Kang P, McAlinden C, Wildsoet CF. Effects of multifocal soft contact lenses used to slow myopia progression on quality of vision in young adults. Acta Ophthalmol. 2017 Feb;95(1):e43-e53. doi: 10.1111/aos.13173. Epub 2016 Aug 6. PMID 27495880
- [Background] Kim E, Bakaraju RC, Ehrmann K. Power Profiles of Commercial Multifocal Soft Contact Lenses. Optom Vis Sci. 2017 Feb;94(2):183-196. doi: 10.1097/OPX.0000000000000998. PMID 27748699
- [Background] Li SM, Kang MT, Wu SS, Meng B, Sun YY, Wei SF, Liu L, Peng X, Chen Z, Zhang F, Wang N. Studies using concentric ring bifocal and peripheral add multifocal contact lenses to slow myopia progression in school-aged children: a meta-analysis. Ophthalmic Physiol Opt. 2017 Jan;37(1):51-59. doi: 10.1111/opo.12332. Epub 2016 Nov 23. PMID 27880992
- [Background] Liu Y, Wildsoet C. The effect of two-zone concentric bifocal spectacle lenses on refractive error development and eye growth in young chicks. Invest Ophthalmol Vis Sci. 2011 Feb 22;52(2):1078-86. doi: 10.1167/iovs.10-5716. Print 2011 Feb. PMID 20861487
- [Background] Liu Y, Wildsoet C. The effective add inherent in 2-zone negative lenses inhibits eye growth in myopic young chicks. Invest Ophthalmol Vis Sci. 2012 Jul 31;53(8):5085-93. doi: 10.1167/iovs.12-9628. PMID 22761258
- [Background] Lopes-Ferreira D, Fernandes P, Queiros A, Gonzalez-Meijome JM. Combined Effect of Ocular and Multifocal Contact Lens Induced Aberrations on Visual Performance: Center-Distance Versus Center-Near Design. Eye Contact Lens. 2018 Sep;44 Suppl 1:S131-S137. doi: 10.1097/ICL.0000000000000355. PMID 28060146
- [Background] McFadden SA, Tse DY, Bowrey HE, Leotta AJ, Lam CS, Wildsoet CF, To CH. Integration of defocus by dual power Fresnel lenses inhibits myopia in the mammalian eye. Invest Ophthalmol Vis Sci. 2014 Feb 14;55(2):908-17. doi: 10.1167/iovs.13-11724. PMID 24398103
- [Background] Sankaridurg P. Contact lenses to slow progression of myopia. Clin Exp Optom. 2017 Sep;100(5):432-437. doi: 10.1111/cxo.12584. Epub 2017 Jul 28. PMID 28752898
- [Background] Smith EL 3rd, Kee CS, Ramamirtham R, Qiao-Grider Y, Hung LF. Peripheral vision can influence eye growth and refractive development in infant monkeys. Invest Ophthalmol Vis Sci. 2005 Nov;46(11):3965-72. doi: 10.1167/iovs.05-0445. PMID 16249469
- [Background] Smith EL 3rd, Hung LF, Huang J, Arumugam B. Effects of local myopic defocus on refractive development in monkeys. Optom Vis Sci. 2013 Nov;90(11):1176-86. doi: 10.1097/OPX.0000000000000038. PMID 24061154
- [Background] Tarrant J, Severson H, Wildsoet CF. Accommodation in emmetropic and myopic young adults wearing bifocal soft contact lenses. Ophthalmic Physiol Opt. 2008 Jan;28(1):62-72. doi: 10.1111/j.1475-1313.2007.00529.x. PMID 18201337
- [Background] Tse DY, To CH. Graded competing regional myopic and hyperopic defocus produce summated emmetropization set points in chick. Invest Ophthalmol Vis Sci. 2011 Oct 17;52(11):8056-62. doi: 10.1167/iovs.10-5207. PMID 21911586
- [Background] Walline JJ, Lindsley K, Vedula SS, Cotter SA, Mutti DO, Twelker JD. Interventions to slow progression of myopia in children. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD004916. doi: 10.1002/14651858.CD004916.pub3. PMID 22161388
- [Background] Walline JJ, Greiner KL, McVey ME, Jones-Jordan LA. Multifocal contact lens myopia control. Optom Vis Sci. 2013 Nov;90(11):1207-14. doi: 10.1097/OPX.0000000000000036. PMID 24061152
- [Background] Wallman J, Wildsoet C, Xu A, Gottlieb MD, Nickla DL, Marran L, Krebs W, Christensen AM. Moving the retina: choroidal modulation of refractive state. Vision Res. 1995 Jan;35(1):37-50. doi: 10.1016/0042-6989(94)e0049-q. PMID 7839608